CLINICAL TRIAL: NCT06964347
Title: A Randomized Clinical Trial Comparing the Analgesic Efficacy of Combined Local Anesthetic Blockade and Neuromodulation (Hybrid Technique) Versus Local Anesthetic Blockade Only for Analgesia After Below-knee Amputation
Brief Title: Combined Local Anesthetic Blockade and Neuromodulation vs Local Anesthetic Blockade Only for Analgesia After Below-knee Amputation: RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chi-Ho Ban Tsui, Professor-Med Ctr Line, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 73646
Record Dates: First submitted 2024-01-09; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Amputation
Keywords: peripheral nerve stimulation; neuromodulation; peripheral nerve block; post-amputation pain; below-knee amputation

STUDY DESIGN:
Intervention Model Description: Comparison of two groups: 1) Group Hybrid block 2) Group LA block
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study team members collecting the data and participating subjects will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group Hybrid block (Experimental): Continuous local anesthetic infusion through the nerve block catheter and peripheral nerve stimulation.
  Interventions: Device: Ropivacaine 0.2% + nerve stimulator set
- Group LA block (Active Comparator): Continuous local anesthetic infusion through the nerve block catheter.
  Interventions: Drug: Ropivacaine 0.2%

INTERVENTIONS:
Device: Ropivacaine 0.2% + nerve stimulator set — Patients will receive a continuous local anesthetic (LA) infusion through the popliteal sciatic nerve block catheter using an infusion of ropivacaine 0.2% at a rate of 8-12 ml/h for at least 3 postoperative days. In addition, patients will receive a low-frequency peripheral nerve stimulation (PNS) via a nerve stimulator set to the pre-determined setting of adequate clinical response (determined in the preoperative area).
  Arms: Group Hybrid block
Drug: Ropivacaine 0.2% — Patients will receive a continuous local anesthetic infusion through the popliteal sciatic nerve block catheter using an infusion of ropivacaine 0.2% at a rate of 8-12 ml/h for at least 3 postoperative days. In addition, patients will have an inactive PNS button for the purposes of blinding.
  Arms: Group LA block

SUMMARY:
This multi-site clinical trial aims to assess the efficacy and safety of combining peripheral nerve stimulation with local anesthetic nerve blockade compared to the standard of care, i.e., local anesthetic blockade only using safe stimulation parameters in a condition associated with high postoperative pain state, i.e. a patient undergoing lower limb amputation.

DETAILED DESCRIPTION:
The primary aim of this pilot trial is to evaluate the feasibility, safety, and analgesic efficacy of the hybrid technique (combined PNS and LA-based PNB) compared to that of PNB during the hospital course in patients undergoing below-knee amputations. The secondary aims are to estimate analgesia and opioid-sparing effects at later timepoints of 3, 6, and 12 months following the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age
* Undergoing below-knee amputation

Exclusion Criteria:

* Chronic opioid use (daily use within the two weeks before surgery and duration of use of more than four weeks of > 30 mg of oxycodone per day or > 50 of morphine milligrams per day)
* Neuromuscular deficit of the target nerve(s)
* Compromised immune system or concurrent risk of infection based on medical history (e.g., immunosuppressive therapies such as chemotherapy, radiation, sepsis, infection).
* Implanted spinal cord stimulator, cardiac pacemaker/defibrillator, deep brain stimulator, or another implantable neurostimulator whose stimulus current pathway may overlap
* History of bleeding disorder or chronic antiplatelet or anticoagulation therapies (other than aspirin) that require to be restarted within the first three postoperative days
* Allergy to study medications or devices (including occlusive dressings, bandages, tape, etc.)
* Incarceration
* Pregnancy
* Chronic pain for more than three months of any severity in an anatomic location other than the surgical site
* Anxiety disorder
* History of substance abuse
* Inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pain scores | First 24 postoperative hours
  Decrease in the proportional incidence of severe or intolerable pain scores (11-point numerical rating scale (NRS) from 0-10, 0 signifying no pain, 10 signifying the worse pain)

SECONDARY OUTCOMES:
Analgesic consumption | At 24, 48, and 72 postoperative hours
  Cumulative rescue and breakthrough analgesic consumption
Quality of recovery (QoR-15) | At postoperative clinic visit (around 1-2 weeks)
  Survey based on patient-reported outcomes. There are 15 questions based on a scale of 0-10, 0 signifying the worst outcome, 10 signifying the best, for a score range of 0-150.
Pain scores | At 12 hour time intervals over the 72 hours
  Static and dynamic pain scores (11-point numerical rating scale (NRS) from 0-10, 0 signifying no pain, 10 signifying the worse pain)
Brief Pain Inventory - short form | During the preoperative assessment and at the 3 and 6 months postoperative assessments.
  A self-reported scale that assesses both the severity of pain and impact of pain on daily functioning, each question assessed on an 11-point scale, where 0 represents the best outcome and 10 - the worst outcome. The score range is 0-110.
Phantom limb pain | At 1 week, three months, 6 months and 1 year
  The incidence of phantom limb and residual limb pain in both groups
Adverse events | Duration of postoperative recovery (typically 1-2 weeks)
  Block and opioid-related adverse events
Time to ambulation | Duration of postoperative recovery (typically 1-2 weeks)
  Number of post-operative days until ambulation
Hospital length of stay | Duration of postoperative recovery (typically 1-2 weeks)
  Number of post-operative days spent in hospital

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Stanford University, Stanford, California
  - Mayo Clinic, Jacksonville, Florida
  - University of Iowa, Iowa City, Iowa
- University of Alberta, Edmonton, Canada

IPD SHARING:
Plan to Share IPD: No